CLINICAL TRIAL: NCT02226744
Title: Focused Breathing Study
Brief Title: Study to Measure Relaxation From Different Types of Focused Breathing Exercises
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No funds to complete study as anticipated, preliminary data used for future grant
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Gurjeet Birdee, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 131700
Record Dates: First submitted 2014-08-20; First posted 2014-08-27 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Breathing; Mind-body Practices; Yoga; Meditation
Keywords: breathing; mind-body practices; yoga; meditation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Focused breathing (Active Comparator): Focused deep breathing techniques used to produce specific physiological and psychological states
  Interventions: Behavioral: Focused Breathing
- Focused breathing 2 (Active Comparator): Focused deep breathing techniques used to produce specific physiological and psychological states
  Interventions: Behavioral: Focused Breathing

INTERVENTIONS:
Behavioral: Focused Breathing

SUMMARY:
Mind-body practices, such as yoga, ta'i chi, mindfulness and biofeedback, commonly use slow breathing techniques to induce physiological and mental relaxation. Medical research suggests that slow breathing techniques induce physiological relaxation. This 6 week study will compare the effects of different types of breathing. The hypothesis is that different breathing techniques produce different physiological and mental changes.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 50 years
* English speaking

Exclusion Criteria:

* Hypertension
* Heart disease: history of coronary artery disease, myocardial infarction, significant valvular disease, or congestive heart failure
* Diabetes
* Renal Disease
* Anxiety Disorder
* Depression
* Other psychiatric conditions including schizophrenia or bipolar disorder
* Attention-deficit-disorder or Attention-deficit-hyperactivity disorder
* Musculoskeletal condition limiting capacity to perform yoga such as chronic lower back pain, chronic neck pain
* Asthma
* Chronic Obstructive Lung Disease
* Obstructive Sleep Apnea
* Smoker
* Currently taking blood pressure medications, oral diabetic medication or insulin
* Current participation in a mind-body practice/program
* Current cancer other than non-melanoma skin cancer
* Regular swimmer
* Plays wind or brass musical instruments

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Magnitude of changes in heart rate response to upright position | 10 minutes at baseline, 2 weeks and 6 weeks

SECONDARY OUTCOMES:
Magnitude of changes in heart rate variability measured as ratio of low frequency to high frequency ratio components (Hz) | Baseline, 2 weeks, and 6 weeks
Magnitude of changes in catecholamines in response to upright position | 10 minutes at baseline, 2 weeks, and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gurjeet S Birdee, MD MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States